CLINICAL TRIAL: NCT03201458
Title: A Randomized Phase 2 Study of Atezolizumab in Combination With Cobimetinib Versus Atezolizumab Monotherapy in Participants With Unresectable Cholangiocarcinoma
Brief Title: Atezolizumab With or Without Cobimetinib in Treating Patients With Metastatic Bile Duct Cancer That Cannot Be Removed by Surgery or Gallbladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2017-01127; NCI-2017-01127 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ETCTN10139; 10139 (Other: JHU Sidney Kimmel Comprehensive Cancer Center LAO); 10139 (Other: CTEP); UM1CA186691 (NIH)
Record Dates: First submitted 2017-06-27; First posted 2017-06-28 (Actual); Results first posted 2023-07-11 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-02

CONDITIONS: Gallbladder Carcinoma; Metastatic Cholangiocarcinoma; Stage III Intrahepatic Cholangiocarcinoma AJCC v8; Stage IV Intrahepatic Cholangiocarcinoma AJCC v8; Unresectable Cholangiocarcinoma
MeSH Terms: conditions — Gallbladder Neoplasms; Cholangiocarcinoma | interventions — atezolizumab; Biopsy; Specimen Handling; cobimetinib; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (atezolizumab) (Experimental): Patients receive atezolizumab IV over 30-60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI and collection of blood samples throughout the trial and undergo tumor biopsy on study.
  Interventions: Drug: Atezolizumab; Procedure: Biopsy; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging
- Arm B (atezolizumab, cobimetinib) (Experimental): Patients receive atezolizumab IV over 30-60 minutes on days 1 and 15 and cobimetinib PO QD on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI and collection of blood samples throughout the trial and undergo tumor biopsy on study.
  Interventions: Drug: Atezolizumab; Procedure: Biopsy; Procedure: Biospecimen Collection; Drug: Cobimetinib; Procedure: Computed Tomography; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Procedure: Biopsy — Undergo tumor biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cobimetinib — Given PO
  Other Names: Cotellic; GDC-0973; MEK Inhibitor GDC-0973; XL518
  Arms: Arm B (atezolizumab, cobimetinib)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; tomography
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI

SUMMARY:
This randomized phase II trial studies how well atezolizumab with or without cobimetinib works in treating patients with bile duct cancer that has spread to other places in the body (metastatic) and cannot be removed by surgery (unresectable) or gallbladder cancer. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Cobimetinib is used in patients whose cancer has a mutated (changed) form of a gene called BRAF. It is in a class of medications called kinase inhibitors. It works by blocking the action of an abnormal protein that signals cancer cells to multiply. This helps slow or stop the spread of cancer cells. Giving atezolizumab with cobimetinib may work better at treating patients with bile duct and gallbladder cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the progression free survival (PFS) of patients receiving atezolizumab monotherapy and cobimetinib in combination with atezolizumab for unresectable cholangiocarcinoma.

SECONDARY OBJECTIVES:

I. To assess the overall survival (OS) of patients receiving cobimetinib in combination with atezolizumab and atezolizumab monotherapy for unresectable cholangiocarcinoma.

II. To determine the objective response rate (ORR), defined as complete plus partial response, of cobimetinib in combination with atezolizumab and atezolizumab monotherapy in patients with unresectable cholangiocarcinoma.

III. To assess the safety and tolerability of cobimetinib in combination with atezolizumab and atezolizumab monotherapy in patients with unresectable cholangiocarcinoma.

IV. To determine the relationship between PD-L1 expression in tumor at baseline and on treatment, and response to treatment.

CORRELATIVE OBJECTIVES:

I. To determine the effect of cobimetinib on CD8+ T cell infiltration in tumor. II. To determine the effect of cobimetinib on T cell subpopulations systemically and in tumor, PD-1/PD-L1 expression on tumor, and MHC 1/2 expression.

III. To determine the effect of cobimetinib on markers of immune exhaustion and pro-apoptotic factors in CD8+ effector T cells.

IV. To explore the effect of cobimetinib on local and systemic immune activation pathways and immune suppressive pathways through expression profiling.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive atezolizumab intravenously (IV) over 30-60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) or magnetic resonance imaging (MRI) and collection of blood samples throughout the trial and undergo tumor biopsy on study.

ARM B: Patients receive atezolizumab IV over 30-60 minutes on days 1 and 15 and cobimetinib orally (PO) once daily (QD) on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo CT or MRI and collection of blood samples throughout the trial and undergo tumor biopsy on study.

After completion of study treatment, patients are followed up every 3 months until death, withdrawal of consent, or study closure, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed metastatic or unresectable cholangiocarcinoma or gallbladder carcinoma (GBC), having received at least 1 prior line of systemic therapy, and received no more than 2 prior lines of therapy in the metastatic setting (disease recurrence =< 6 months from the last dose of adjuvant therapy in resected patients will be considered the first line of therapy)

  * Includes intrahepatic cholangiocarcinoma (IHC), extrahepatic cholangiocarcinoma (EHC), and gallbladder carcinoma (GBC), but not ampulla of vater cancers
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) with conventional techniques or as >= 10 mm (>= 1 cm) with spiral CT scan, MRI, or calipers by clinical exam; assessment must be completed within 4 weeks of randomization
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of cobimetinib in combination with atezolizumab in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 80%)
* Life expectancy of greater than 2 months
* Leukocytes >= 2,500/mcL (within 2 weeks of randomization)
* Absolute neutrophil count >= 1,500/mcL (within 2 weeks of randomization)
* Platelets >= 75,000/mcL (within 2 weeks of randomization)
* Hemoglobin >= 8 g/dL (within 2 weeks of randomization)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (however, patients with known Gilbert disease who have serum bilirubin level =< 3 x ULN may be enrolled) (within 2 weeks of randomization)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x ULN (within 2 weeks of randomization)
* Creatinine clearance >= 30 mL/min/1.73 m^2 by Cockcroft-Gault OR creatinine < 1.5 x ULN (within 2 weeks of randomization)
* International normalized ratio (INR) and activated partial thromboplastin time (aPTT) =< 1.5 x ULN (this applies only to patients who do not receive therapeutic anticoagulation; patients receiving therapeutic anticoagulation, such as low-molecular-weight heparin or warfarin, should be on a stable dose) (within 2 weeks of randomization)
* Administration of atezolizumab and cobimetinib may have an adverse effect on pregnancy and poses a risk to the human fetus, including embryo-lethality; women of childbearing potential must agree to use either two adequate barrier methods or a barrier method plus a hormonal method of contraception to prevent pregnancy, or to abstain from heterosexual activity (complete abstinence) prior to study entry, for the duration of study participation, and for 5 months (150 days) after the last dose of study agent; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; male patients must agree to use an adequate method of contraception, or to abstain from heterosexual activity (complete abstinence), prior to study entry, for the duration of study participation, and for 5 months (150 days) after the last dose of study agent
* Ability to understand and the willingness to sign a written informed consent document
* Patients positive for human immunodeficiency virus (HIV) are allowed on study, but HIV-positive patients must have:

  * A stable regimen of highly active anti-retroviral therapy (HAART)
  * No requirement for concurrent antibiotics or antifungal agents for the prevention of opportunistic infections
  * A CD4 count above 250 cells/mcL and an undetectable HIV viral load on standard polymerase chain reaction (PCR)-based tests
* Oxygen saturation >= 92% on room air

Exclusion Criteria:

* Received chemotherapy or radiotherapy within 3 weeks prior to randomization or those who have not recovered to =< grade 1 adverse events (other than alopecia) due to agents administered more than 3 weeks earlier; herbal therapy intended as anticancer therapy must be discontinued at least 1 week prior to randomization; for patients who received prior immunotherapy (eg anti-CTLA-4), at least five drug half-lives must have passed before the patient may enroll on this study; however, the following therapies are allowed:

  * Hormone-replacement therapy or oral contraceptives
  * Palliative radiotherapy for bone metastases >= 2 weeks prior to randomization
* Prior treatment with a MEK inhibitor or ERK inhibitor
* Prior treatment with any anti-PD-1 or anti-PD-L1 antibody, prior allogeneic bone marrow transplantation, or prior solid organ transplantation
* Treatment with any investigational agent within 4 weeks prior to cycle 1, day 1, or five drug half-lives (whichever is longer)
* Treatment with systemic immunosuppressive medications (including, but not limited to, prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 6 weeks prior to cycle 1 day 1;

  * Patients who have received acute, low dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled
  * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
* Patients with known primary central nervous system (CNS) malignancy or symptomatic CNS metastases, with the following exceptions:

  * Patients with asymptomatic treated CNS metastases may be enrolled, provided all the criteria listed above are met as well as the following:

    * Radiographic demonstration of clinical stability upon the completion of CNS directed therapy and no evidence of interim progression between the completion of CNS directed therapy and the screening radiographic study
    * No stereotactic radiation or whole-brain radiation within 28 days prior to randomization
    * Screening CNS radiographic study >= 4 weeks from completion of radiotherapy and >= 2 weeks from discontinuation of corticosteroids
* Has a known concurrent malignancy that is expected to require active treatment within two years, or may interfere with the interpretation of the efficacy and safety outcomes of this study in the opinion of the treating investigator; superficial bladder cancer, non-melanoma skin cancers, or low grade prostate cancer not requiring therapy should not exclude participation in this trial
* Known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Allergy or hypersensitivity to components of the cobimetinib formulations
* History of congenital long QT syndrome or corrected QT interval (QTc) > 450 msec within 2 weeks of randomization
* Left ventricular ejection fraction (LVEF) below institutional lower limit of normal (LLN) or below 50%, whichever is lower, as determined by echocardiogram or multi-gated acquisition (MUGA) scan within 4 weeks of randomization
* Patients who meet any of the following exclusion criteria related to ocular disease will be excluded from study entry:

  * Known risk factors for ocular toxicity, consisting of any of the following:

    * History of serous retinopathy
    * History of retinal vein occlusion (RVO)
    * Evidence of ongoing serous retinopathy or RVO at screening
* Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 enzymes are ineligible; these include St. John's wort or hyperforin (potent CYP3A4 enzyme inducer) and grapefruit juice (potent cytochrome P450 CYP3A4 enzyme inhibitor); such substances can significantly increase or decrease the serum level of cobimetinib; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; fatty liver; and inherited liver disease

  * Patients with past or resolved hepatitis B infection (defined as having a negative hepatitis B surface antigen [HBsAg] test and a positive anti-HBc [antibody to hepatitis B core antigen] antibody test) are eligible
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV ribonucleic acid (RNA)
* History or risk of autoimmune disease, including, but not limited to, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Bell's palsy, Guillain-Barre syndrome, multiple sclerosis, autoimmune thyroid disease, vasculitis, or glomerulonephritis

  * Patients with a history of autoimmune hypothyroidism on a stable dose of thyroid replacement hormone may be eligible
  * Patients with controlled type 1 diabetes mellitus on a stable insulin regimen may be eligible
  * Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

    * Rash must cover less than 10% of body surface area (BSA)
    * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, flucinolone 0.01%, desonide 0.05%, aclometasone dipropionate 0.05%)
    * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan; history of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Severe infections within 4 weeks prior to randomization, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of infection within 2 weeks prior to randomization
* Received oral or intravenous (IV) antibiotics within 2 weeks prior to randomization; patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or chronic obstructive pulmonary disease) are eligible
* Major surgical procedure within 4 weeks prior to randomization or anticipation of need for a major surgical procedure during the course of the study
* Administration of a live, attenuated vaccine within 4 weeks before randomization or anticipation that such a live, attenuated vaccine will be required during the study and up to 5 months after the last dose of atezolizumab

  * Influenza vaccination should be given during influenza season only (approximately October to March); patients must not receive live, attenuated influenza vaccine within 4 weeks prior to cycle 1, day 1 or at any time during the study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, active tuberculosis (TB), symptomatic congestive heart failure (CHF), unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

  * Symptomatic CHF is defined as New York Heart Association (NYHA) CHF class II or higher disease
* Pregnant women are excluded from this study because both atezolizumab and cobimetinib are expected to cause fetal harm if used during pregnancy; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with cobimetinib or atezolizumab, breastfeeding should be discontinued if the mother is treated with either therapy; these potential risks may also apply to other agents used in this study
* Inability or unwillingness to swallow pills
* History of malabsorption syndrome or other condition that would interfere with enteral absorption
* Clinically significant ascites, defined as ascites that is symptomatic or has resulted in a paracentesis in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2020-08-07 (Actual); Study Completion 2024-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nilofer S Azad, Principal Investigator — JHU Sidney Kimmel Comprehensive Cancer Center LAO
Locations (41):
- United States (41):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope South Pasadena, South Pasadena, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Derived] Yarchoan M, Cope L, Ruggieri AN, Anders RA, Noonan AM, Goff LW, Goyal L, Lacy J, Li D, Patel AK, He AR, Abou-Alfa GK, Spencer K, Kim EJ, Davis SL, McRee AJ, Kunk PR, Goyal S, Liu Y, Dennison L, Xavier S, Mohan AA, Zhu Q, Wang-Gillam A, Poklepovic A, Chen HX, Sharon E, Lesinski GB, Azad NS. Multicenter randomized phase II trial of atezolizumab with or without cobimetinib in biliary tract cancers. J Clin Invest. 2021 Dec 15;131(24):e152670. doi: 10.1172/JCI152670. PMID 34907910

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A (Atezolizumab): Patients receive atezolizumab IV over 30-60 minutes on days 1 and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
- Arm B (Atezolizumab, Cobimetinib): Patients receive atezolizumab IV over 30-60 minutes on days 1 and 15 and cobimetinib PO QD on days 1-21. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm A (Atezolizumab) | Arm B (Atezolizumab, Cobimetinib)
Started | 43 | 43
Completed | 39 | 38
Not Completed | 4 | 5
Not completed — No longer eligible | 2 | 5
Not completed — Health event before starting | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Atezolizumab) | Arm B (Atezolizumab, Cobimetinib) | Total
Number analyzed (Participants) | 43 | 43 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 4 | 5
  Between 18 and 65 years | 32 | 28 | 60
  >=65 years | 10 | 11 | 21
Age, Continuous [Median (Full Range); unit: years] | 62 [45 to 86] | 63 [44 to 80] | 63 [44 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 23 | 53
  Male | 13 | 20 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 8 | 12
  Not Hispanic or Latino | 39 | 33 | 72
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 33 | 37 | 70
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 43 | 43 | 86
Subgroup [Count of Participants; unit: Participants]
  Extrahepatic cholangiocarcinoma (EHC) | 9 | 9 | 18
  Gallbladder cancer (GBC) | 12 | 10 | 22
  Intrahepatic cholangiocarcinoma (IHC) | 22 | 24 | 46
Height [Median (Full Range); unit: centimeter (cm)] | 163.4 [142.2 to 190.0] | 166.4 [151.0 to 182.9] | 164.9 [142.2 to 190.0]
Weight [Median (Full Range); unit: kilogram (kg)] | 71.5 [44.0 to 151.3] | 78.5 [38.3 to 121.9] | 76.9 [38.3 to 151.3]
Body Surface Area [Median (Full Range); unit: meters squared (m^2)] | 1.81 [1.39 to 2.83] | 1.90 [1.27 to 2.29] | 1.89 [1.27 to 2.83]

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS within each treatment arm will be summarized descriptively and compared between groups, under the assumption of Cox proportional hazards, using the stratified log-rank test to account for tumor site. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From date of randomization to time of progression or death, assessed up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Atezolizumab) | Arm B (Atezolizumab, Cobimetinib)
Number analyzed (Participants) | 39 | 38
Participants
  Progression free at 1 Year after Randomization | 0 | 3
  Progressed or Off Treatment by 1 Year after Randomization | 39 | 35
Statistical Analysis 1: Comparison: Arm A (Atezolizumab) vs Arm B (Atezolizumab, Cobimetinib); Test type: Superiority; p = 0.027, Log Rank — One-sided test; Hazard Ratio (HR) = 0.58, 90% CI 2-sided [0.35 to 0.93]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Will be assessed using National Cancer Institute's Common Terminology Criteria for Adverse Events version 5.0. The incidence of AEs will be tabulated by subgroups of interest (e.g. grade 3 or higher, organ class, relationship to study drug). For analyses at the individual level, the highest grade and relationship to study drug will be assumed if multiple events have occurred. Toxicity will be tabulated by type and grade and will be summarized with descriptive statistics.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Atezolizumab) | Arm B (Atezolizumab, Cobimetinib)
Number analyzed (Participants) | 39 | 38
Participants
  Grade 3 or higher adverse event considered at least possibly related to the study drug(s) | 15 | 17
  No grade 3 or higher adverse events considered at least possibly related to the study drug(s) | 24 | 21
Statistical Analysis 1: Comparison: Arm A (Atezolizumab) vs Arm B (Atezolizumab, Cobimetinib); Test type: Superiority; p = 0.22, Fisher Exact; Odds Ratio (OR) = 2.3

3. Secondary Outcome: Objective Response Rate
Description: Defined as the proportion of response evaluable subjects who have a complete response or partial response and will be assessed by Response Evaluation Criteria in Solid Tumors version 1.1. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 1 year
Population: Evaluable population excluded patients removed from study prior to the first radiographic evaluation time point for clinical progression or death from tumor progression.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Atezolizumab) | Arm B (Atezolizumab, Cobimetinib)
Number analyzed (Participants) | 36 | 30
Participants
  Complete Response | 0 | 0
  Partial Response | 1 | 1
  Stable Disease | 10 | 13
  Clinical or Radiographic Progression | 25 | 16

4. Secondary Outcome: Overall Survival
Description: Results will be summarized descriptively and compared between groups, under the assumption of proportional hazards, using the stratified log-rank test to account for tumor site.
Time Frame: From date of randomization to time of death, assessed up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Atezolizumab) | Arm B (Atezolizumab, Cobimetinib)
Number analyzed (Participants) | 39 | 38
Participants
  Alive at 1 year | 9 | 9
  Deceased or Lost to Follow Up at 1 year | 30 | 29
Statistical Analysis 1: Comparison: Arm A (Atezolizumab) vs Arm B (Atezolizumab, Cobimetinib); Test type: Superiority; p = 0.410, Log Rank — One-sided test

5. Secondary Outcome: Change in CD8+ Density Within the Tumor
Description: Change between the pre-treatment tumor biopsy to the on-treatment biopsy collected on day 21.
Time Frame: Day 21
Population: Participants with paired high-quality biopsies (fold change pre- and post-treatment).
Measure: Mean (Standard Deviation); unit: cells per millimeter squared
Arm/Group | Arm A (Atezolizumab) | Arm B (Atezolizumab, Cobimetinib)
Number analyzed (Participants) | 8 | 5
cells per millimeter squared | 0.719 (0.469) | 0.892 (0.535)

6. Other Pre Specified Outcome: Number of Participants With PD-L1 Expression
Description: The number of participants with tumors expressing PD-L1 by 1 percent or more.
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Atezolizumab) | Arm B (Atezolizumab, Cobimetinib)
Number analyzed (Participants) | 9 | 9
Participants
  1% or more Positivity | 1 | 1
  No expression | 8 | 8

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Arm A (Atezolizumab) | Arm B (Atezolizumab, Cobimetinib)
All-Cause Mortality (participants affected / at risk) | 35/43 | 35/43
Serious Adverse Events (participants affected / at risk) | 32/43 | 31/43
Other Adverse Events (participants affected / at risk) | 38/43 | 36/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Atezolizumab) (N=43) | Arm B (Atezolizumab, Cobimetinib) (N=43)
Abdominal distention (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 6 | 4
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Altered mental status (Psychiatric disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 2
Ascites (Gastrointestinal disorders) | 0 | 5
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Bacteremia (Infections and infestations) | 1 | 0
Biliary duct obstruction (Hepatobiliary disorders) | 1 | 4
Biliary tract infection (Infections and infestations) | 1 | 0
Blood bilirubin increased (Investigations) | 2 | 1
Cardiac troponin increased (Investigations) | 1 | 0
Chills (General disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 2 | 3
Colonic obstruction (Gastrointestinal disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 3
Duodenal obstruction (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Edema limbs (General disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 2
Esophagitis (Gastrointestinal disorders) | 0 | 1
Facial muscle weakness (Nervous system disorders) | 0 | 1
Fatigue (General disorders) | 1 | 3
Fever (General disorders) | 0 | 5
Bone fracture (Injury, poisoning and procedural complications) | 0 | 1
Fungemia (Infections and infestations) | 1 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 4 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Ileal obstruction (Gastrointestinal disorders) | 1 | 0
Infusion related reaction (General disorders) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Malaise (General disorders) | 0 | 1
Meningitis (Infections and infestations) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 2
Gastric obstruction (Gastrointestinal disorders) | 2 | 0
Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Peritoneal infection (Infections and infestations) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 0 | 3
Presyncope (Nervous system disorders) | 1 | 0
Sepsis (Infections and infestations) | 1 | 5
Sinus tachycardia (Cardiac disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Small intestinal perforation (Gastrointestinal disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 1
Herpes zoster (Skin and subcutaneous tissue disorders) | 0 | 1
Ureteral obstruction (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 2
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Vasovagal reaction (Nervous system disorders) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 5
Disease Progression (General disorders) | 32 | 31
Stroke (Nervous system disorders) | 0 | 1
Death NOS (General disorders) | 2 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Atezolizumab) (N=43) | Arm B (Atezolizumab, Cobimetinib) (N=43)
Abdominal distension (Gastrointestinal disorders) | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 14 | 15
Alanine aminotransferase (ALT) increased (Investigations) | 10 | 9
Alkaline phosphatase increased (Investigations) | 12 | 17
Allergic reaction (Immune system disorders) | 3 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Anemia (Blood and lymphatic system disorders) | 13 | 16
Anorexia (Metabolism and nutrition disorders) | 9 | 7
Anxiety (Psychiatric disorders) | 2 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Ascites (Gastrointestinal disorders) | 4 | 4
Aspartate aminotransferase (AST) increased (Investigations) | 15 | 14
Atrial fibrillation (Cardiac disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Belching (Gastrointestinal disorders) | 0 | 2
Bloating (Gastrointestinal disorders) | 5 | 3
Blood bilirubin increased (Investigations) | 7 | 3
Chills (General disorders) | 5 | 4
Constipation (Gastrointestinal disorders) | 7 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 5
Creatinine increased (Investigations) | 6 | 3
Creatinine kinase (CK) increased (Investigations) | 0 | 9
Dehyrdation (Metabolism and nutrition disorders) | 5 | 4
Diarrhea (Gastrointestinal disorders) | 14 | 23
Dizziness (Nervous system disorders) | 4 | 7
Dry eye (Eye disorders) | 0 | 2
Dry mouth (Gastrointestinal disorders) | 1 | 7
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 3
Dysgeusia (Nervous system disorders) | 2 | 3
Dyspepsia (Gastrointestinal disorders) | 3 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 9
Edema (General disorders) | 4 | 16
Fatigue (General disorders) | 20 | 24
Fever (General disorders) | 9 | 13
Flatulence (Gastrointestinal disorders) | 2 | 4
Gastroesophageal reflux disease (GERD) (Gastrointestinal disorders) | 1 | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 4
Headache (Nervous system disorders) | 4 | 4
Hematuria (Renal and urinary disorders) | 0 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 3 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 12
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 4
Hypertension (Vascular disorders) | 13 | 9
Hypoalbuminemia (Metabolism and nutrition disorders) | 11 | 19
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 7
Hypokalemia (Metabolism and nutrition disorders) | 11 | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 5 | 6
Hyponatremia (Metabolism and nutrition disorders) | 12 | 12
Hypophosphotemia (Metabolism and nutrition disorders) | 3 | 3
Hypotension (Vascular disorders) | 2 | 0
Hypothyroidism (Endocrine disorders) | 4 | 3
Infusion-related reaction (General disorders) | 4 | 2
Insomnia (Psychiatric disorders) | 2 | 5
Lipase increased (Investigations) | 1 | 4
Lymphocyte count decreased (Investigations) | 13 | 17
Malaise (General disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Nausea (Gastrointestinal disorders) | 12 | 17
Neutrophil count decreased (Investigations) | 3 | 4
Non-cardiac chest pain (General disorders) | 2 | 0
Oral pain (Gastrointestinal disorders) | 2 | 0
Pain (General disorders) | 8 | 9
Peripheral neuropathy (Nervous system disorders) | 2 | 4
Platelet count decreased (Investigations) | 9 | 21
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Proteinuria (Renal and urinary disorders) | 2 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 9
Rash (Skin and subcutaneous tissue disorders) | 4 | 30
Sinus bradycardia (Cardiac disorders) | 1 | 2
Sinus tachycardia (Cardiac disorders) | 2 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Thrush (Infections and infestations) | 3 | 0
Vomiting (Gastrointestinal disorders) | 10 | 18
Weight loss (Investigations) | 5 | 2
White blood cell decreased (Investigations) | 7 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT03201458/Prot_SAP_000.pdf